CLINICAL TRIAL: NCT03265197
Title: Evaluation of Adding Lidocaine to Dexamethasone in Intra-tympanic Injection for Management of Tinnitus
Acronym: tinnitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: saad elzayat (Other)
Responsible Party: Sponsor-Investigator, saad elzayat, doctor and lecturer of ORL, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KafrelsheikhU
Record Dates: First submitted 2016-07-05; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Tinnitus
Keywords: Tinnitus; Intra-tympanic; Lidocaine; Dexamethasone
MeSH Terms: conditions — Tinnitus | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intratympanic injection of drugs; (Experimental): intervention by Intratympanic injection of drugs in two studied groups; group A, injection of combined 2 drugs( lidocaine and dexamethasone) and group B, injection of one drug (dexamethasone only).
  Interventions: Drug: Intra-tympanic injection of drugs
- Data management of Intratympanic drugs (Active Comparator): intervention by Manage data of two study group as blind statistical between group A, injection of combined 2 drugs( lidocaine and dexamethasone) and group B, injection of one drug (dexamethasone only).
  Interventions: Other: Data management of intratympanic drugs

INTERVENTIONS:
Drug: Intra-tympanic injection of drugs — Intratympanic injection of combined lidocaine and dexamethasone in treatment of tinnitus
  Other Names: Lidocaine in tinnitus
  Arms: Intratympanic injection of drugs;
Other: Data management of intratympanic drugs — intervention by statistical analysis of Intratympanic injection of combined lidocaine and dexamethasone in treatment of tinnitus
  Arms: Data management of Intratympanic drugs

SUMMARY:
Importance; Tinnitus is a heterogeneous diagnosis that may occur alone, in the presence of hearing loss or as a component of other disorders and can be quite disabling. Intratympanic injections of medications recently proved to have role in management of tinnitus. The investigators report on our experience with the use of intratympanic injection of Lidocaine as local anesthetic which potentiate the action of dexthamesasone in treatment of tinnitus without adding potential risks of inner ear Objective; to describe the effect of Lidocaine as local anesthetic may potentiate the action of dexthamesasone intratympanic injection in treatment of tinnitus without adding potential risks of inner ear Design, Setting, participants ; For this single tertiary center( Tanta University Hospital ) prospective case series, the investigators included 44 patients divided into two groups (A and B) 22 patients in each group suffering from tinnitus between March 2015 and October 2015 Intervention; Under local anesthesia 22 patients were subjected to intratympanic injection with combined Lidocaine 2% and dexamethasone with ratio (1:1), in the group A, and 22 patients in the other group B were subjected to intratympanic injection with dexamethasone only , this process was repeated 3 times for 3 successive weeks.

Main Outcome and Measures; the primary outcome is self-reported significant improve in tinnitus in group A more in group B without adding significant damage of inner ear

DETAILED DESCRIPTION:
Introduction Tinnitus is a heterogeneous diagnosis that may occur alone, in the presence of hearing loss, or as a component of other disorders and can be quite disabling. Tinnitus has been estimated to affect over 10% of population.1 Attempts to treat and classify tinnitus date back to ancient Egypt. The Ebers Papyrus includes great detail regarding the "treatment for a bewitched ear'' Infusion of medicine into the ear were common at this time. (2500 BC).2 It is more prevalent in patients between the ages of 50 and 70 years, with men over 65 years being afflicted more often than women of similar age. 3-4 Tinnitus has complex pathophysiology which is difficult to understand and investigate. Many studies have indicated that, it usually occurs due to redirection of information and the role of the non-classical auditory pathways, changes in synaptic efficacy can open connections in the CNS that are normally not conducting and that can redirect information in the CNS. 5 Subjective tinnitus is conscious perception of phantom sound, which is audible by the patients only and affects their routine life. Many therapies and drugs have been used in the treatment of tinnitus, such as dietary modification, tinnitus retraining therapy, antidepressants, anxiolytics, and herbal medicines. However, no significant improvement has been found in the majority of the patients treated by these therapies or drugs. Various attempts have been made to treat peripheral tinnitus since the 1940s, by way of intra tympanic injection. This administration procedure requires only low concentrations of medication and comes with minimal systemic exposure thus avoiding serious systemic side effects. 6 Intra-tympanic treatment of tinnitus with Lidocaine, Corticosteroids and\or Aminoglycosides has been used to treat disabling symptoms of tinnitus with different results. 7 Intra-tympanic drug perfusion, has been successively used to treat tinnitus since the 1990s.4 Lidocaine (Xylocaine), also called lignocaine, is a potent local anesthetic agent, widely used both topical and injection anesthesia. The mechanism of action of Lidocaine on the auditory system in the subjective tinnitus is controversial as it has central and peripheral action. 7 Therefore, this study was designed in a prospective randomized controlled fashion to evaluate the efficacy and safety of adding Lidocaine to dexamethasone in treatment of idiopathic subjective tinnitus.

Methods:

Trial Designs Two identical, prospective, double-blind controlled Single center randomized clinical trials assessed the effectiveness, safety, and tolerability of adding Lidocaine to dexamethasone in intratympanic injection in patients with idiopathic subjective tinnitus (age range 30 to 63 years). The study design and consent forms were approved by the research ethics committee of Tanta university hospitals. The study was conducted according to the Declaration of Helsinki and a written informed consent was obtained from every patient who agreed to participate in the study.

The study was carried out on 44 patients suffering from prominent unilateral idiopathic subjective non-pulsatile tinnitus (IST) attending to the outpatient clinic of otorhinolaryngology department of the Tanta University Hospital, from March 2015 to October 2015. They were 18 male and 26 female, with age ranged from 30 to 63 years old (mean 48.909±7.758). Patients were equally divided into two groups (A and B). Group A was injected by combined Lidocaine 2% and dexamethasone 8mg/2ml. Group B was injected only by dexamethasone 8mg/2ml. Exclusion criteria included Extreme age, pulsatile tinnitus, objective tinnitus and ear inflammation.

Randomization and Trial Intervention Every patient was given a code number in the study to keep his personal information confidential. Adequate provisions to maintain privacy of participants and confidentiality of data were taken into consideration. To avoid selection bias, each candidate, who signed an informed consent for participation in the study, was given a number from one to forty four. For every two consecutive patients; the first was enrolled in group A and the second was enrolled in group B till the end of the 44 patients.

Operative technique The drum was anaesthetized locally by cotton soaked with Xylocaine 10%. The patient was kept in supine position and his head turned about 45°away from the surgeon. All patients were injected by a single surgeon (dr saad elzayat,MD, consultant of ORL). The assigned solution was injected under direct vision through an operating microscope at the anterosuperior quadrant of the tympanic membrane using a 27-gauge needle. About one ml of the drug was injected in the diseased ear. In group A, the investigators used combined Lidocaine 2% and dexamethasone (8mg/2ml) with ratio (1:1). In group B, the investigators used dexamethasone only for injection 8mg/2ml. The patients would remain in the supine position for about 30 minutes and avoid swallowing after the injection to keep the Eustachian tube closed and give the drug maximal time of contact with the round window. The patients were kept in our department for six hours for observation of any complications. This procedure was repeated for three times at weekly interval.

Follow up visits were scheduled one month, 3 months and six months from the first injection. Before and after injection, each patient was asked to complete Tinnitus Handicap Inventory (THI) and Tinnitus Functional Index (TFI) questionnaires. Full otological, audiological examination and adverse events were recorded.

Statistical Analysis Sample size was calculated as 22 patients in each group to give the study a power of 80% at the 5% level of significance. At the time of randomization and during the follow up period, both the patient and the surgeon were unaware of the group assignment. Each patient was coded; these codes were kept with the main investigator. The envelope was opened on the day of the operation. During the follow up period, the patient was assigned to the principal investigator of the thesis. The study sheet summarized all the information related to the patient except the operative data. The sheet was copied and added to the patient file after each session, whereas the original sheet was kept in the study folder. Statistical presentation and analysis of the present study was conducted, using SPSS V17. Chicago IL, SPSS Inc®)

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic subjective non-pulsatile tinnitus (IST)

Exclusion Criteria:

* Extreme age, pulsatile tinnitus, objective tinnitus and ear inflammation.

Ages: 30 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
measuring tinnitus scales improvements by using dexmethsone alone and by using combined lidocaine and tinnitus | 6 months
  using measuring indice as Tinnitus Handicap Inventory (THI)self-perceived tinnitus handicap severity.
measuring medication complication and side effect by using hearing test indicators | 6 months
  using hearing indices as pure tone audiometry (PTA) ,

IPD SHARING:
Plan to Share IPD: Yes
publication in ORL journal

REFERENCES:
- [Background] Adams PF, Hendershot GE, Marano MA; Centers for Disease Control and Prevention/National Center for Health Statistics. Current estimates from the National Health Interview Survey, 1996. Vital Health Stat 10. 1999 Oct;(200):1-203. PMID 15782448
- [Background] She W, Dai Y, Du X, Chen F, Ding X, Cui X. Treatment of subjective tinnitus: a comparative clinical study of intratympanic steroid injection vs. oral carbamazepine. Med Sci Monit. 2009 Jun;15(6):PI35-9. PMID 19478715
- [Background] Moller AR. Pathophysiology of tinnitus. Otolaryngol Clin North Am. 2003 Apr;36(2):249-66, v-vi. doi: 10.1016/s0030-6665(02)00170-6. PMID 12856295
- [Background] Meyer T. Intratympanic treatment for tinnitus: a review. Noise Health. 2013 Mar-Apr;15(63):83-90. doi: 10.4103/1463-1741.110285. PMID 23571297
- [Background] Elzayat S, El-Sherif H, Hegazy H, Gabr T, El-Tahan AR. Tinnitus: Evaluation of Intratympanic Injection of Combined Lidocaine and Corticosteroids. ORL J Otorhinolaryngol Relat Spec. 2016;78(3):159-66. doi: 10.1159/000445774. Epub 2016 Jun 1. PMID 27245783
- [Result] Dodson KM, Sismanis A. Intratympanic perfusion for the treatment of tinnitus. Otolaryngol Clin North Am. 2004 Oct;37(5):991-1000. doi: 10.1016/j.otc.2004.03.003. PMID 15474106